CLINICAL TRIAL: NCT03340740
Title: The Effect of Cetirizine on Bronchoconstriction in Patients With Allergic Rhinitis and Wheezing in the Pediatric Emergency Department
Brief Title: The Effect of Cetirizine on Bronchoconstriction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Stephen M. Blumberg, Primary Investigator, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-8047
Record Dates: First submitted 2017-10-04; First posted 2017-11-13 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Allergic Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic; Asthma | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The medication and placebo doses will be prepared in the pharmacy at the study site and provided to the investigators in deidentified bottles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cetirizine (Experimental): Cetirizine 10mg (10ml) (patients age 12-17) or cetirizine 5mg (5ml) (patients age 6-11) x 1 dose at beginning of course in emergency department.
  Interventions: Drug: Cetirizine Hydrochloride 1 MG/ML
- Placebo (Placebo Comparator): Placebo 10ml (patients age 12-17) or 5ml (patients age 6-11) x 1 dose at beginning of course in the emergency department.
  Interventions: Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: Cetirizine Hydrochloride 1 MG/ML — Cetirizine oral suspension
  Arms: Cetirizine
Drug: Placebo - Concentrate — Similar-appearing liquid to cetirizine oral suspension
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of cetirizine, an oral antihistamine, on wheezing in patients with allergic rhinitis. Patients presenting to the pediatric emergency department who have a history of allergic rhinitis and who are wheezing will be asked to participate. Half of patients will receive a dose of cetirizine and the other half will receive placebo and their response will be monitored over the course of their emergency department visit with vital signs, physical examinations, and measurement of bronchoconstriction with spirometry.

DETAILED DESCRIPTION:
This is a prospective randomized, placebo-controlled trial to look at the effect of cetirizine on bronchoconstriction in patients with allergic rhinitis who present to the Pediatric Emergency Department with wheezing. Oral second generation antihistamines such as cetirizine are already the standard of care for allergic rhinitis. Wheezing pediatric patients with allergic rhinitis who are not already on this therapy will be randomized to receive either age-appropriate-dosed cetirizine or placebo in addition to standard asthma therapy at the discretion of the treating clinician, and will be monitored every 30 minutes with asthma scores and FEV1 measurements. At the conclusion of 3 hours, each patient who received placebo will receive a dose of cetirizine, and each patient who received cetirizine will receive a placebo medication dose, such that initiating therapy for allergic rhinitis is delayed by no more than 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic rhinitis
* Wheezing

Exclusion Criteria:

* Use of antihistamine within the past 72 hours
* Chronic Pulmonary Condition other than asthma
* Other contraindication to cetirizine
* Severe asthma exacerbation requiring resuscitation

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Index Score between baseline and 3 hours | At baseline and at 3 hours
  A composite score on a scale of 0-14, comprised of respiratory rate, wheezing, inspiration/expiration ratio, accessory muscle use and oxygen saturation.

SECONDARY OUTCOMES:
Change in FEV1 between baseline and 3 hours | At baseline and at 3 hours
  FEV 1 will be measured using a commercially-available spirometry device.

OTHER OUTCOMES:
Number of patients admitted to the hospital for inpatient management of wheezing | At 3 hours
  Admission to hospital or discharge home

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Blumberg, MD, Principal Investigator — Jacobi Medical Center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No